CLINICAL TRIAL: NCT06657729
Title: Evaluation of Oral Feeding Skills of Very Premature Infants
Brief Title: Oral Feeding Skills of Very Premature Infants
Acronym: NUTRIO
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0741; 2024-A01791-46 (Other: ID RCB)
Record Dates: First submitted 2024-10-16; First posted 2024-10-24 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Extreme Prematurity (gestational Age Below 29 Weeks)
Keywords: prematurity; orality; sucking; feeding autonomy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Extremely preterm infants: Extremely preterm infants born before 29 weeks.
  Interventions: Other: Succiometry

INTERVENTIONS:
Other: Succiometry — Assessement of sucking performance by measuring pressures (suction, crushing) with a succiometer every 10 days. This instrument consists of a standard silicone teat for premature newborns, which is connected via two silicone tubes to pressure micro-sensors. These pressure sensors measure the child's sucking activity on the teat. This activity is characterised by suction and crushing movements. It is a non-nutritive sucking activity (no fluid is delivered). Sucking performance is recorded during a period of calm awakening of the infant and over a period of 5 minutes, and is part of routine care since non-nutritive sucking is a common practice in neonatal unit. The first measurement will be taken in the first week of life and then every 7-10 days until discharge from the neonatal unit.

SUMMARY:
Extremely premature infants, born at a gestational age (GA) of less than 29 weeks, are exposed to numerous complications in the neonatal period (digestive, cardiac, infectious, respiratory, neurological) and in the longer term (neurosensory and cognitive development, impaired growth, oral feeding disorders). In premature babies, non-nutritive sucking is present from 27 weeks' gestation, but the "suck, swallow, breathe" sequence, which is essential for feeding autonomy, does not mature until 34 weeks, with wide individual variations. Therefore, preterm newborns initially needs a gastric tube to receive enteral nutrition. During this period, the oral sphere is often dys-stimulated by the insertion/attachment of the gastric tube, aspirations of oral secretions, etc. The earlier children are born, the more frequent and serious the pathologies associated with prematurity, the more frequent these dys-stimulations are and the longer enteral feeding via gastric tube is required. As a result, the more immature the child, the more the development of oral performance is disrupted. This disrupts the transition from enteral feeding to oral feeding and therefore the acquisition of autonomous feeding, which is essential if the child is to be able to go out at home. This has an impact on the length of hospitalisation. Individualised developmental care, the current standard of care in neonatology, aims on the one hand to reduce dys-stimulation and on the other hand to offer positive oral stimulation such as non-nutritive sucking and perioral stimulation. Non-nutritive sucking consists of providing the child with a dummy as often and for as long as possible, i.e. as soon as the child is awake. Some departments also use specific and adapted perioral stimulation protocols. For several years, the department of neonatology at the Croix Rousse University Hospital included in care protocols, a protocol for peri-oral stimulation. It begins as soon as the baby is no longer suffering from any major (haemodynamic or respiratory) problems. It is stopped when feeding is active and autonomy has been achieved. It consists of stimulating the perioral and oral area, ideally four times a day, when the child is awake and particularly before meals. Perioral stimulation is performed on the baby's face, then, depending on the baby's reactions, oral stimulation is performed using a cotton bud soaked in milk. When the baby places his tongue in the sucking position and closes his lips, oral feeding can begin.

In a retrospective, single-centre study carried out in neonatology at the Croix Rousse hospital in 163 babies born before 29 weeks' gestation, the investigator calculated that the average corrected GA for the acquisition of feeding autonomy was 38.3 weeks' gestation, with significant inter-individual variability.

The hypothesis is that extremely premature infants already have oral skills very early, then lose them due to the numerous dys-stimulations of the oral sphere during intensive care period. Stimulations of the oral and perioral sphere, implemented early, could make it possible to limit this loss of competence and to observe a physiological evolution of oral skills.

ELIGIBILITY:
Inclusion Criteria:

* Infant born before 29 GA
* Hospitalized in the Croix Rousse neonatology department
* Admitted within the first three days of life

Exclusion Criteria:

* Discharge (transfer) planned within 15 days of birth
* Silicone allergy
* Severe congenital malformation
* Pathology requiring surgery
* Parental refusal

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born before 29 GA (extreme prematurity), hospitalized in the Neonatal unit of Croix Rousse Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-05-17 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Suckling performances | From date of inclusion until the date of discharge from the neonatal unit, assessed up to 5 months
  The pressure variations recorded when the infant has the teat in its mouth are analysed. Various parameters are quantified to assess suckling performances: 1 - the number of suction peaks.
Suckling performances | From date of inclusion until the date of discharge from the neonatal unit, assessed up to 5 months
  The pressure variations recorded when the infant has the teat in its mouth are analysed. Various parameters are quantified to assess suckling performances: 2 - the amplitude of suction peaks.
Suckling performances | From date of inclusion until the date of discharge from the neonatal unit, assessed up to 5 months
  The pressure variations recorded when the infant has the teat in its mouth are analysed. Various parameters are quantified to assess suckling performances: 3 - the timing of suction peaks.
Suckling performances | From date of inclusion until the date of discharge from the neonatal unit, assessed up to 5 months
  The pressure variations recorded when the infant has the teat in its mouth are analysed. Various parameters are quantified to assess suckling performances: 4 - the number of crushing peaks.
Suckling performances | From date of inclusion until the date of discharge from the neonatal unit, assessed up to 5 months
  The pressure variations recorded when the infant has the teat in its mouth are analysed. Various parameters are quantified to assess suckling performances: 5 - the amplitude of crushing peaks.
Suckling performances | From date of inclusion until the date of discharge from the neonatal unit, assessed up to 5 months
  The pressure variations recorded when the infant has the teat in its mouth are analysed. Various parameters are quantified to assess suckling performances: 6 - the timing of crushing peaks.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Croix Rousse, Lyon, France